CLINICAL TRIAL: NCT03982420
Title: The ENROUTE Transcarotid Neuroprotection System (ENROUTE Transcarotid NPS) DW-MRI Evaluation
Acronym: DW-MRI-US
Status: Completed | Type: Observational
Sponsor: Silk Road Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: SRM-2018-01
Record Dates: First submitted 2019-06-06; First posted 2019-06-11 (Actual); Results first posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Carotid Artery Diseases; Carotid Atherosclerosis; Carotid Stenosis; Carotid Artery Plaque; Carotid Disease
MeSH Terms: conditions — Carotid Artery Diseases; Carotid Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Procedure: Transcarotid Revascularization (TCAR) — Carotid revascularization treated with the FDA-cleared ENROUTE Transcarotid NPS in conjunction with the FDA-approved ENROUTE Transcarotid Stent
  Other Names: Carotid Revascularization, Carotid Artery Stenting

SUMMARY:
The goal of this evaluation is to document the incidence of post procedure DW-MRI lesions (relative to baseline) in patients treated with the transcarotid artery revascularization (TCAR) procedure.

DETAILED DESCRIPTION:
This is a prospective, single-arm, multi-center evaluation of patients requiring carotid revascularization who are treated with the FDA-cleared ENROUTE Transcarotid NPS in conjunction with the FDA-approved ENROUTE Transcarotid Stent System. Both the ENROUTE Transcarotid NPS and ENROUTE Transcarotid Stent System have received CE mark and are commercially available in the European Union.

Patients enrolled in this study will have been offered the TCAR intervention as part of standard of care for the treatment of carotid artery stenosis, regardless of whether or not they agree to be in the study. Therefore, the act of participation in this procedure will not be the determining factor in whether or not the patient receives the TCAR treatment. Subject participation means they agree to undergo two additional DW-MRI imaging procedures immediately after the procedure and at 30 days to determine whether there is an increase in new white lesions. Any other procedure other than the active collection of consent and data by the sponsor is standard of care for the treatment of carotid artery stenosis.

These patients will be monitored to document the incidence of post procedure DW-MRI lesions (relative to baseline).

ELIGIBILITY:
Inclusion Criteria:

* Stenosis must be >50% as determined by ultrasound or angiogram1 and the patient has a history of stroke (minor or non-disabling; NIHSS ≤4 or mRS ≤2), TIA and/or amaurosis fugax within 180 days of the procedure ipsilateral to the carotid artery to be stented.
* Stenosis must be >80% as determined by ultrasound or angiogram without any neurological symptoms within the prior 180 days.
* Target vessel must meet diameter requirements for stent (refer to stent IFU for diameter requirements).
* Patient has a discrete lesion located in the internal carotid artery (ICA) with or without involvement of the contiguous common carotid artery (CCA).
* Patient is willing to comply with the protocol requirements and return to the treatment center for all required clinical evaluations.
* Patient must have a life expectancy ≥ 3 years at the time of the index procedure without contingencies related to other medical, surgical or endovascular intervention.
* Patient meets at least one of the surgical high-risk criteria listed in CMS National Coverage Determination (NCD) for Percutaneous Transluminal Angioplasty (20.7)

Exclusion Criteria

* Alternative source of cerebral embolus
* Patient has chronic atrial fibrillation.
* Patient has had any episode of paroxysmal atrial fibrillation within the past 6 months, or history of paroxysmal atrial fibrillation requiring chronic anticoagulation.
* Knowledge of cardiac sources of emboli. e.g. left ventricular aneurysm, intracardiac filling defect, cardiomyopathy, aortic or mitral prosthetic heart valve, calcific aortic stenosis, endocarditis, mitral stenosis, atrial septal defect, atrial septal aneurysm, or left atrial myxoma).
* Recently (<60 days) implanted heart valve (either surgically or endovascularly), which is a known source of emboli as confirmed on echocardiogram.
* Abnormal angiographic findings: ipsilateral intracranial or extracranial arterial stenosis (as determined by angiography or CTA/MRA ≤ 6 months prior to index procedure) greater in severity than the lesion to be treated, cerebral aneurysm > 5 mm, AVM (arteriovenous malformation) of the cerebral vasculature, or other abnormal angiographic findings.
* Patient has a history of spontaneous intracranial hemorrhage within the past 12 months, or has had a recent (<7 days) stroke of sufficient size (on CT or MRI) to place him or her at risk of hemorrhagic conversion during the procedure (less than one-third middle cerebral artery volume).
* Patient had hemorrhagic transformation of an ischemic stroke within the past 60 days.
* Patient with a history of major stroke attributable to either carotid artery (CVA or retinal embolus) with major neurological deficit (NIHSS ≥ 5 OR mRS ≥ 3) likely to confound study endpoints within 1 month of index procedure.
* Patient has an evolving stroke.
* Patient has an intracranial tumor.
* Patient has neurologic illnesses within the past two years characterized by fleeting or fixed neurologic deficit which cannot be distinguished from TIA or stroke, including but not limited to: moderate to severe dementia, partial or secondarily generalized seizures, complicated or classic migraine, tumor or other space-occupying brain lesions, subdural hematoma, cerebral contusion or other post-traumatic lesions, intracranial infection, demyelinating disease, or intracranial hemorrhage).
* Patient has had a TIA or amaurosis fugax within 48 hrs prior to the procedure.
* Patient has an isolated hemisphere defined as the ipsilateral middle cerebral artery being supplied only by the ipsilateral internal carotid artery.
* Patient has active bleeding diathesis or coagulopathy or will refuse blood transfusion.
* Patient had or will have CABG, endovascular stent procedure, valve intervention or vascular surgery within 30 days before or after the intervention.
* Myocardial Infarction within 72 hours prior to the intervention.
* Occlusion of the ipsilateral common or internal carotid artery.
* An intraluminal filling defect (defined as an endoluminal lucency surrounded by contrast, seen in multiple angiographic projections, in the absence of angiographic evidence of calcification) whether or not it is associated with an ulcerated target lesion.
* Patients with carotid string sign (a very high-grade carotid stenosis to the skull base with a long, thin, barely visible string of contrast within the true lumen of the artery.).
* Ostium of Common Carotid Artery (CCA) requires revascularization (>50% stenosis).
* Patient has an open stoma in the neck.
* Patients with hostile necks due to prior neck irradiation
* Female patients who are pregnant
* Patient has history of intolerance or allergic reaction to any of the study medications or stent materials (refer to stent IFU), including aspirin (ASA), ticlopidine, clopidogrel, prasugrel, statin or contrast media (that can't be pre medicated). Patients must be able to tolerate statins and a combination of ASA and ticlopidine, ASA and clopidogrel or ASA and prasugrel.
* Patient has a life expectancy <3 years with contingencies related to other medical, surgical, or interventional procedures as per the Wallaert Score and patients with primary, recurrent or metastatic malignancy who do not have independent assessment of life expectancy performed by the treating oncologist or an appropriate specialist other than the physician performing TCAR.
* Patient has had a recent GI bleed that would interfere with antiplatelet therapy.
* Patient is actively participating in an investigational drug or device trial (IND or IDE) that has not completed the required protocol follow-up period.
* Patient has inability to understand and cooperate with study procedures.
* Presence of extensive or diffuse atherosclerotic disease involving the proximal common carotid artery that would preclude the safe introduction of the study device.
* Patient is otherwise unsuitable for intervention in the opinion of the physician.
* Patients who cannot have MRI due to metallic implants (e.g. orthopedic implants, pacemakers, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients participating in this evaluation will be comprised of male and female symptomatic or asymptomatic patients requiring carotid revascularization.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-01-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (5):
  - Yale University, New Haven, Connecticut
  - Indiana University, Vascular Surgery, Indianapolis, Indiana
  - Newton Wellesley Hospital, Newton, Massachusetts
  - Stony Brook University Medical Center, Stony Brook, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
- Clinica Universidad de Navarra, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Results will be published following study end date.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were considered enrolled after signing the informed consent and having undergone a successful Transcarotid artery revascularization (TCAR) procedure (e.g., the procedure was not aborted due to technical issues or due to local complications that precluded stent implantation). Patients who were screened but did not meet all study criteria were considered screen failures and were not enrolled.
Groups:
- Single-arm: Patients requiring carotid revascularization who were treated with the FDA-cleared ENROUTE Transcarotid NPS in conjunction with the FDA-approved ENROUTE Transcarotid Stent System.
Period: Overall Study
Arm/Group | Single-arm
Started | 55
Completed | 54
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single-arm
Number analyzed (Participants) | 55
Age, Customized [Count of Participants; unit: Participants]
  ≤64 Years Old | 6
  65-69 Years old | 9
  70-74 Years old | 19
  75-79 Years old | 11
  ≥80 Years old | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 4
  Caucasian | 35
  Hispanic or Latino | 15
  Unknown | 1
Height (cm) [Mean (Standard Deviation); unit: CM] | 169.5 (9.63)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 81.9 (13.48)
High Risk Factors [Count of Participants; unit: Participants]
  Contralateral carotid artery occlusion: Yes | 7
  Contralateral carotid artery occlusion: No | 48
  Tandem stenoses >70%: Yes | 2
  Tandem stenoses >70%: No | 53
  High cervical carotid artery stenosis: Yes | 23
  High cervical carotid artery stenosis: No | 32
  Restenosis after carotid endarterectomy: Yes | 11
  Restenosis after carotid endarterectomy: No | 44
  Bilateral carotid artery stenosis requiring treatment: Yes | 0
  Bilateral carotid artery stenosis requiring treatment: No | 55
  Hostile Necks safe for transcarotid access: Yes | 1
  Hostile Necks safe for transcarotid access: No | 54
  Hostile Necks safe for transcarotid access Radical neck dissection: Yes | 2
  Hostile Necks safe for transcarotid access Radical neck dissection: No | 53
  Hostile Necks safe for transcarotid access Cervical spine immobility: Yes | 5
  Hostile Necks safe for transcarotid access Cervical spine immobility: No | 50
  ≥75 years of age: Yes | 21
  ≥75 years of age: No | 34
  ≥2-vessel coronary artery disease and history of angina: Yes | 8
  ≥2-vessel coronary artery disease and history of angina: No | 47
  History of angina, unstable or CCS of 3 or 4: Yes | 2
  History of angina, unstable or CCS of 3 or 4: No | 53
  Congestive heart failure (CHF), NYHA Functional Class III or IV: Yes | 2
  Congestive heart failure (CHF), NYHA Functional Class III or IV: No | 53
  Severe left ventricular dysfunction: LVEF <30%: Yes | 0
  Severe left ventricular dysfunction: LVEF <30%: No | 55
  Myocardial infarction >72 hours and <6 weeks prior to the procedure: Yes | 0
  Myocardial infarction >72 hours and <6 weeks prior to the procedure: No | 55
  Severe pulmonary disease (COPD): Yes | 3
  Severe pulmonary disease (COPD): No | 52
  Permanent contralateral cranial nerve injury: Yes | 1
  Permanent contralateral cranial nerve injury: No | 54
  Patient has chronic renal insufficiency: Yes | 2
  Patient has chronic renal insufficiency: No | 53
Subjects with Multiple High-Risk Criteria. Number of High-Risk Factors [Count of Participants; unit: Participants]
  0 High-Risk Factors | 0
  1 High-Risk Factors | 30
  2 High-Risk Factors | 18
  3 or More High-Risk Factors | 7

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Ipsilateral New White Lesions, by Patient
Description: Number of Participants with new white lesions from baseline (pre-procedure) by Diffusion-Weighted Magnetic Resonance Imaging (DW-MRI) between 12-60 hours after procedure end time up to 30 days post-procedure.
Time Frame: Between 12-60 hours after procedure end time to 30 days post-procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Single-arm
Number analyzed (Participants) | 55
Participants | 12

2. Primary Outcome: Incidence of Ipsilateral Persistent Lesions, by Patient
Description: Number of participants at 30 day post-procedure with persistent ipsilateral new white lesions post-procedure by Diffusion-Weighted Magnetic Resonance Imaging (DW-MRI).
Time Frame: 30-days
Population: 3 patients did not complete the 30-day DW-MRI.
Measure: Count of Participants; unit: Participants
Arm/Group | Single-arm
Number analyzed (Participants) | 52
Participants | 3

3. Secondary Outcome: All Stroke and Neurological Death
Description: Number of Participants who experienced Stroke or Neurological death between 12-60 hours after procedure end time up to 30 days post-procedure.
Time Frame: 0 to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Single-arm
Number analyzed (Participants) | 55
Participants
  Stroke: Yes | 0
  Stroke: No | 55
  Neurological Death: Yes | 0
  Neurological Death: No | 55

4. Secondary Outcome: Volume of DW-MRI White Lesions
Description: Volume of Persistent new white lesions post-procedure by Diffusion-Weighted Magnetic Resonance Imaging (DW-MRI) at 30-Days.
Time Frame: 30-days
Population: Out of the 55 subjects who participated in this study, 3 participants had a total of 5 persistence white lesions at 30 days. The volume relates to the number of persistent white lesions (5).
Measure: Mean (Full Range); unit: Cubic Centimeter (cc)
Units Other Than Participants: Persistent White Lesions
Arm/Group | Single-arm
Number analyzed (Participants) | 3
Number analyzed (Persistent White Lesions) | 5
Cubic Centimeter (cc) | 0.21 [0.02 to 0.98]

5. Secondary Outcome: Location of DW-MRI Lesions
Description: Number persistent new white lesions post-procedure by location by Diffusion-Weighted Magnetic Resonance Imaging (DW-MRI) at 30-Days, categorized by location.
Time Frame: 30-day
Population: Out of the 55 subjects who participated in this study, 3 participants had a total of 5 persistence white lesions located in the Middle Cerebral Artery at 30 days.
Measure: Number; unit: Lesion
Units Other Than Participants: Persistent White Lesions
Arm/Group | Single-arm
Number analyzed (Participants) | 3
Number analyzed (Persistent White Lesions) | 5
Lesion
  Middle Cerebral Artery (MCA) Territory - Persistent 30-day lesion | 5
  Posterior Cerebral Artery (PCA) Territory - Persistent 30-day lesion | 0
  Anterior Cerebral Artery (ACA) Territory - Persistent 30-day lesion | 0

6. Secondary Outcome: Stroke/Neurological Death in Patients Eligible and Ineligible for ROADSTER 2
Description: No patients enrolled in this study were enrolled in ROADSTER 2 trial; therefore, ROADSTER 2 specific endpoints were not evaluated.
Time Frame: 0 to 30-day
Population: None of the patients enrolled in this study were enrolled in ROADSTER 2 study. Therefore, ROADSTER 2 specific endpoints were not evaluated.
Arm/Group | Single-arm
Number analyzed (Participants) | 0

7. Secondary Outcome: Rate of Contralateral New White Lesions by Diffusion-Weighted Magnetic Resonance Imaging (DW-MRI), by Patient
Description: Subjects with persistent contralateral new white lesions post-procedure by Diffusion-Weighted Magnetic Resonance Imaging (DW-MRI), at 30-Days.
Time Frame: 30-day
Measure: Count of Participants; unit: Participants
Arm/Group | Single-arm
Number analyzed (Participants) | 55
Participants | 0

ADVERSE EVENTS:
Time Frame: Post-Procedure to 30-day
Arm/Group | Single-arm
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55
Other Adverse Events (participants affected / at risk) | 0/55

LIMITATIONS AND CAVEATS:
Modest sample size. Not powered for formal hypothesis testing or subgroup comparisons. No comparator arm with CEA or TF-CAS to enabled direct comparisons. Variability in contrast injection technique may influence lesion detection. Power injection was recommended but not universally followed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI's right to publish individual results is restricted until after the multi-center publication is complete. The sponsor also reserves the right to review and approve all publications or presentations prior to submission.

DOCUMENTS (1):
  • Study Protocol (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/20/NCT03982420/Prot_000.pdf